CLINICAL TRIAL: NCT06763848
Title: Protein A Immunoadsorption for the Treatment of Acute Episodes of Neuromyelitis Optica Spectrum Disorder：A Multicenter, Open-label, Superiority, Randomised Trial
Brief Title: Protein A immuNoaDsorption for the Treatment of Acute Episodes of Neuromyelitis Optica Spectrum Disorder
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other); Guangdong 999 Brain Hospital (Other); Second Xiangya Hospital of Central South University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wei Qiu, Chief Physician, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-330-02; WQiu (Registry Identifier: WQiu)
Record Dates: First submitted 2024-12-15; First posted 2025-01-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
Keywords: neuromyelitis optica spectrum disorders; immunoadsorption; acute episodes; treatment
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): The experimental group was treated with a combination of protein A immunoadsorption and intravenous methylprednisolone. The methylprednisolone was administered following a regimen of 1g for 5 days, 0.5g for 3 days, 0.25g for 2 days, and 0.12g for 1 day. Protein A immunoadsorption was conducted every other day, unless a physician determined that the patient's condition was unsuitable for treatment, in which case treatment was administered according to medical advice. A total of 5 treatments were given, with each session involving the regeneration of plasma at 1 to 3 times the plasma volume. Sequentially, the patients in this group were uniformly administered oral immunosuppressants, specifically azathioprine or mycophenolate mofetil (MMF).
  Interventions: Device: Protein A immunoadsorption
- control group (Active Comparator): The control group was treated with intravenous methylprednisolone, following a regimen of 1g for 5 days, 0.5g for 3 days, 0.25g for 2 days, and 0.12g for 1 day.Sequentially, the patients in this group were uniformly administered oral immunosuppressants, specifically azathioprine or mycophenolate mofetil (MMF).
  Interventions: Drug: intravenous methylprednisolone

INTERVENTIONS:
Device: Protein A immunoadsorption — The experimental group was treated with a combination of protein A immunoadsorption and intravenous methylprednisolone. The methylprednisolone was administered following a regimen of 1g for 5 days, 0.5g for 3 days, 0.25g for 2 days, and 0.12g for 1 day. Protein A immunoadsorption was conducted every other day, unless a physician determined that the patient's condition was unsuitable for treatment, in which case treatment was administered according to medical advice. A total of 5 treatments were given, with each session involving the regeneration of plasma at 1 to 3 times the plasma volume.
  Arms: experimental group
Drug: intravenous methylprednisolone — The control group was treated with intravenous methylprednisolone, following a regimen of 1g for 5 days, 0.5g for 3 days, 0.25g for 2 days, and 0.12g for 1 day.
  Arms: control group

SUMMARY:
To clarify the efficacy and safety of protein A immunoadsorption therapy for acute exacerbations of neuromyelitis optica spectrum disorders(NMOSD), we designed a multicenter, open-label, superiority randomized controlled clinical trial, planning to enroll 144 patients with NMOSD. We plan to treat patients with acute NMOSD using protein A immunoadsorption combined with high-dose intravenous methylprednisolone, and compare this with treatment using high-dose intravenous methylprednisolone alone. The aim is to observe the impact and safety of protein A immunoadsorption on the treatment efficacy for these patients experiencing acute exacerbations of NMOSD, ultimately providing more comprehensive clinical evidence to support treatment protocols for the acute phase of NMOSD.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study are as follows:

  1. clinical diagnosis of acute Neuromyelitis Optica Spectrum Disorders (NMOSD)
  2. Age and Gender: Participants must be between 18 and 65 years old, inclusive, with no gender restrictions.
  3. Serological Marker: Participants must test positive for AQP4-IgG using the cell-based assay (CBA) method.
  4. Understanding and Consent: Participants or their legal representatives must be able to understand the study's purpose, demonstrate sufficient compliance with the study protocol, and sign the informed consent form.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Participants who cannot establish peripheral or central venous access, or have a history of allergic reactions to plasmapheresis.
3. Participants with contraindications to intravenous methylprednisolone treatment.
4. Participants who have used monoclonal antibodies in the last 6 months, or FcRn antagonists in the last 3 months.
5. Participants who must use ACE inhibitors (ACEI) within 1 week before the start of treatment or during the study, and cannot discontinue their use.
6. Severe Bleeding or Bleeding Disorders
7. Severe Heart Failure
8. Severe Infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of the treatment, the change in the Kurtzke Expanded Disability Status Scale (EDSS) score is evaluated one month after the start of treatment compared to the baseline. The baseline is defined as the patient's condition before | Evaluation timing includes from the screening period to the baseline and the EDSS score assessment one month after starting treatment.
  To assess the effectiveness of the treatment, the change in the Kurtzke Expanded Disability Status Scale (EDSS) score is evaluated one month after the start of treatment compared to the baseline. The baseline is defined as the patient's condition before treatment began, or if the patient had not yet reached a plateau during the initial treatment phase and continued to worsen during hospitalization, the most severe stage during the current hospitalization is used as the baseline.The EDSS is a scale used for the objective and repeatable quantification of disability in patients, with scores ranging from 0 to 10. A score of 0 indicates normal function, while a score of 10 indicates death. An increase in the EDSS score reflects worsening symptoms.The method of evaluation involves calculating the EDSS score difference as follows:
  EDSS Score Difference = EDSS Score (Baseline) - EDSS Score (1 Month After Treatment Start).

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Wang J, Li C, Liu X, Chu M, Chang Y, Wang Y, Wang X, Yu B, Ling L, Yang H, Yang H, Hu X, Qiu W. Rescue immunoadsorption treatment for neuromyelitis optica spectrum disorder attacks unresponsive to intravenous methylprednisolone. J Neuroimmunol. 2021 Jul 15;356:577604. doi: 10.1016/j.jneuroim.2021.577604. Epub 2021 May 7. PMID 33992860
- [Background] Kleiter I, Gahlen A, Borisow N, Fischer K, Wernecke KD, Wegner B, Hellwig K, Pache F, Ruprecht K, Havla J, Krumbholz M, Kumpfel T, Aktas O, Hartung HP, Ringelstein M, Geis C, Kleinschnitz C, Berthele A, Hemmer B, Angstwurm K, Stellmann JP, Schuster S, Stangel M, Lauda F, Tumani H, Mayer C, Zeltner L, Ziemann U, Linker R, Schwab M, Marziniak M, Then Bergh F, Hofstadt-van Oy U, Neuhaus O, Winkelmann A, Marouf W, Faiss J, Wildemann B, Paul F, Jarius S, Trebst C; Neuromyelitis Optica Study Group. Neuromyelitis optica: Evaluation of 871 attacks and 1,153 treatment courses. Ann Neurol. 2016 Feb;79(2):206-16. doi: 10.1002/ana.24554. Epub 2015 Nov 26. PMID 26537743
- [Background] Kleiter I, Gahlen A, Borisow N, Fischer K, Wernecke KD, Hellwig K, Pache F, Ruprecht K, Havla J, Kumpfel T, Aktas O, Hartung HP, Ringelstein M, Geis C, Kleinschnitz C, Berthele A, Hemmer B, Angstwurm K, Stellmann JP, Schuster S, Stangel M, Lauda F, Tumani H, Mayer C, Krumbholz M, Zeltner L, Ziemann U, Linker R, Schwab M, Marziniak M, Then Bergh F, Hofstadt-van Oy U, Neuhaus O, Zettl UK, Faiss J, Wildemann B, Paul F, Jarius S, Trebst C; NEMOS (Neuromyelitis Optica Study Group). Apheresis therapies for NMOSD attacks: A retrospective study of 207 therapeutic interventions. Neurol Neuroimmunol Neuroinflamm. 2018 Sep 26;5(6):e504. doi: 10.1212/NXI.0000000000000504. eCollection 2018 Nov. PMID 30345331
- [Background] Trebst C, Jarius S, Berthele A, Paul F, Schippling S, Wildemann B, Borisow N, Kleiter I, Aktas O, Kumpfel T; Neuromyelitis Optica Study Group (NEMOS). Update on the diagnosis and treatment of neuromyelitis optica: recommendations of the Neuromyelitis Optica Study Group (NEMOS). J Neurol. 2014 Jan;261(1):1-16. doi: 10.1007/s00415-013-7169-7. Epub 2013 Nov 23. PMID 24272588
- [Background] Lennon VA, Wingerchuk DM, Kryzer TJ, Pittock SJ, Lucchinetti CF, Fujihara K, Nakashima I, Weinshenker BG. A serum autoantibody marker of neuromyelitis optica: distinction from multiple sclerosis. Lancet. 2004 Dec 11-17;364(9451):2106-12. doi: 10.1016/S0140-6736(04)17551-X. PMID 15589308
- [Background] Wingerchuk DM, Banwell B, Bennett JL, Cabre P, Carroll W, Chitnis T, de Seze J, Fujihara K, Greenberg B, Jacob A, Jarius S, Lana-Peixoto M, Levy M, Simon JH, Tenembaum S, Traboulsee AL, Waters P, Wellik KE, Weinshenker BG; International Panel for NMO Diagnosis. International consensus diagnostic criteria for neuromyelitis optica spectrum disorders. Neurology. 2015 Jul 14;85(2):177-89. doi: 10.1212/WNL.0000000000001729. Epub 2015 Jun 19. PMID 26092914